CLINICAL TRIAL: NCT07029360
Title: Adjunctive Use of Coenzyme Q10 and Probiotics to Improve Periodontal Health in Pregnant Women: A Randomized Controlled Trial
Brief Title: Effectiveness of Coenzyme Q10 and Probiotics in Periodontal Therapy During Pregnancy
Acronym: PREG-Q10
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-Q10PROBIOPREG
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy; Periodontal Disease; Gingivitis; Dental Plaque; Probiotics; Coenzyme Q10; Microbiota
Keywords: Bleeding on Probing; Clinical Attachment Loss; Coenzyme Q10; Dental Plaque; Gingival Inflammation; Gingivitis; Limosilactobacillus reuteri; Microbiota; Non-Surgical Periodontal Treatment; Oral Microbiota; Periodontal Therapy; Plaque Control; Plaque Index; Pregnancy; Pregnant Women; Probiotics; Randomized Controlled Trial
MeSH Terms: conditions — Periodontal Diseases; Gingivitis; Dental Plaque

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Coenzyme Q10 Plus Probiotics (Experimental): Participants assigned to this arm will undergo professional oral hygiene every three months and will follow a home-care regimen consisting of twice-daily use of a coenzyme Q10-based toothpaste combined with a daily probiotic supplement (Limosilactobacillus reuteri Prodentis®, 1 tablet per day) for 6 months. Additional hygiene tools include soft picks and a sonic toothbrush.
  Interventions: Dietary Supplement: Limosilactobacillus reuteri Prodentis®; Other: Coenzyme Q10 Toothpaste
- Coenzyme Q10 Only (Active Comparator): Participants assigned to this arm will undergo professional oral hygiene every three months and will follow a home-care regimen consisting of twice-daily use of a coenzyme Q10-based toothpaste for 6 months, without probiotics. Additional hygiene tools include soft picks and a sonic toothbrush.
  Interventions: Other: Coenzyme Q10 Toothpaste

INTERVENTIONS:
Dietary Supplement: Limosilactobacillus reuteri Prodentis® — Daily administration of Limosilactobacillus reuteri Prodentis® (1 oral tablet per day, taken after brushing in the evening), as an adjunct to non-surgical periodontal therapy and standard home care. Administered for 6 months only in the experimental arm.
  Arms: Coenzyme Q10 Plus Probiotics
Other: Coenzyme Q10 Toothpaste — Twice-daily use of a commercially available toothpaste containing coenzyme Q10, used as part of a home oral hygiene regimen for 6 months. All participants in both study arms will use the same toothpaste, with or without adjunctive probiotic supplementation.

SUMMARY:
This randomized controlled clinical trial aims to evaluate the effectiveness of adjunctive coenzyme Q10 and probiotic supplementation (Limosilactobacillus reuteri Prodentis®) in improving periodontal health in pregnant women undergoing non-surgical periodontal therapy. Forty participants will be randomly assigned to two groups: the test group will receive professional oral hygiene every three months along with a coenzyme Q10-based toothpaste and daily probiotic supplementation; the control group will follow the same protocol without probiotics. The primary outcome is the reduction of the Plaque Index (PI), while secondary outcomes include Bleeding on Probing (BoP), Probing Pocket Depth (PPD), Clinical Attachment Level (CAL), gingival inflammation (MGI, PMGI), plaque distribution (PCR%, API), and gingival recession (R). The study duration is 6 months. The goal is to assess whether this combined therapy can promote a balanced oral microbiota and enhance periodontal health during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between the 4th and 8th month of gestation
* Age ≥ 18 years
* Able to understand and communicate in Italian and/or English
* Willing to provide written informed consent
* Good compliance and willingness to follow study instructions

Exclusion Criteria:

* Presence of cardiac pacemakers
* Diagnosed psychological, neurological, or psychiatric disorders
* Ongoing oncological therapy
* Use of bisphosphonates within the last 12 months
* Poor motivation or low compliance
* Substance abuse (drugs or alcohol) or lifestyle incompatible with study requirements

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only individuals who self-identify as female and are biologically pregnant are eligible to participate in the study.
Enrollment: 40 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-05-15 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Change in Dental Plaque Measured by the Plaque Index Score | Baseline (T0), 1 Month (T1), 3 Months (T2), and 6 Months (T3)
  The Plaque Index (PI) Score will be recorded at four timepoints (baseline, 1 month, 3 months, and 6 months) to assess the amount of dental plaque accumulation. The primary endpoint is the change in PI from baseline (T0) to 6 months (T3), comparing the intervention group (coenzyme Q10 + probiotics) to the control group (coenzyme Q10 only). The index is measured by visually scoring the plaque on tooth surfaces using standardized criteria.
  The Plaque Index score ranges from 0 (no plaque) to 3 (abundant plaque), with higher scores indicating a worse outcome.

SECONDARY OUTCOMES:
Change in Gingival Bleeding Measured by the Bleeding on Probing (BoP) Index | Baseline (T0), 1 Month (T1), 3 Months (T2), and 6 Months (T3)
  The BoP index will be recorded to evaluate gingival bleeding. Comparison will be made between the test group (coenzyme Q10 + probiotics) and the control group (Q10 only) across all study timepoints, from baseline to 6 months. The BoP index is expressed as the percentage of bleeding sites out of the total number of sites examined (range: 0% to 100%), with higher percentages indicating a worse outcome.
Change in Periodontal Pocket Depth Measured by the Probing Pocket Depth (PPD) | Baseline (T0), 1 Month (T1), 3 Months (T2), and 6 Months (T3)
  PPD will be recorded in millimeters to assess periodontal pocket depth. Values will be compared between groups across timepoints to evaluate treatment efficacy. PPD values range from 1 mm (healthy sulcus) to over 7 mm (advanced periodontal disease); higher values indicate a worse outcome.
Change in Clinical Attachment Level Measured by CAL | Baseline (T0), 1 Month (T1), 3 Months (T2), and 6 Months (T3)
  CAL will be measured to assess periodontal tissue support. The difference in attachment level from baseline to 6 months will be analyzed between study groups. CAL is measured in millimeters, typically ranging from 0 mm (no attachment loss) to over 10 mm in severe cases; higher values indicate a worse outcome.
Change in Gingival Inflammation Measured by the Modified Gingival Index (MGI) | Baseline (T0), 1 Month (T1), 3 Months (T2), and 6 Months (T3)
  The MGI will be used to evaluate gingival inflammation. Score changes from baseline to 6 months will be analyzed between the intervention and control groups. The MGI ranges from 0 (normal gingiva) to 4 (severe inflammation), with higher scores indicating a worse outcome.
Change in Interproximal Plaque Measured by the Approximal Plaque Index (API) | Baseline (T0), 1 Month (T1), 3 Months (T2), and 6 Months (T3)
  The API will be used to assess the presence of plaque in interproximal areas. Changes in API scores will be compared between groups over the course of the study. The API is expressed as the percentage of interproximal sites with visible plaque (range: 0% to 100%), with higher values indicating a worse outcome.
Change in Plaque Distribution Measured by Plaque Control Record (PCR%) | Baseline (T0), 1 Month (T1), 3 Months (T2), and 6 Months (T3)
  The PCR% will measure the percentage of oral surfaces with plaque. The effect of the interventions on PCR% will be evaluated from baseline to 6 months. PCR% ranges from 0% (no plaque detected) to 100% (plaque present on all assessed surfaces), with higher values indicating a worse outcome.
Change in Gingival Inflammation Measured by the Papillary Marginal Gingival Index (PMGI) | Baseline (T0), 1 Month (T1), 3 Months (T2), and 6 Months (T3)
  The PMGI will be used to assess inflammation at the gingival margin and papilla. Differences in scores will be analyzed between groups at each follow-up. The PMGI ranges from 0 (normal gingiva) to 5 (severe inflammation with spontaneous bleeding), with higher scores indicating a worse outcome.
Change in Gingival Recession Measured by Clinical Examination | Baseline (T0), 1 Month (T1), 3 Months (T2), and 6 Months (T3)
  Gingival recession (R) will be clinically measured in millimeters to assess changes in gingival margin levels from baseline to 6 months, comparing both groups. Values typically range from 0 mm (no recession) to over 5 mm in severe cases, with higher values indicating a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, Associate Professor, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the corresponding authors.